CLINICAL TRIAL: NCT07248735
Title: Effects of Constraint Induced Movement Therapy With and Without Robotic Glove on Dexterity and Hand Grip Strength in Children With Hemiplegic Cerebral Palsy
Brief Title: Effects of CIMT With and Without Robotic Gloves in Children With Hemiplegic CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/AFTAB ANSAR LODHI
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Child Development Disorder
Keywords: CIMT, Robotic Gloves, Dexterity, Hemiplegic CP
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: This study investigates the impact of CIMT, with and without robotic gloves, on hand dexterity and grip strength in children with hemiplegic CP, aiming to enhance motor skills and promote independence in daily activities. Conducted as a randomized controlled trial at DHQ Hospital, Mandi Bahauddin, the study involves two groups of children aged 6-12 with hemiplegic CP. One group of 17 children will receive CIMT alone with standard treatment, while the other 17 will receive CIMT combined with robotic glove assistance. The robotic glove device aids in flexion, extension, and individual finger movements, providing support for both isolated and coordinated finger actions. Each therapy session will last six hours and be held three to five days a week over four to eight weeks
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Experimental group
  Interventions: Other: CIMT with robotic glove
- Group B (Active Comparator): Control group
  Interventions: Other: CIMT with standard rehabilitation

INTERVENTIONS:
Other: CIMT with robotic glove — The Experimental group undergoes a comprehensive rehabilitation program, combining Constraint-Induced Movement Therapy (CIMT) with robotic glove therapy. The unaffected limb is restrained by the help of Slings, Simple glove, splint or plaster. Each session lasts 6 Hours, occurring 3-5 Days a weekly, over a period of 4-8 weeks. This intensive regimen aims to enhance hand function and mobility by constraining the unaffected hand while using the robotic glove to facilitate precise finger movements.
  Arms: Group A
Other: CIMT with standard rehabilitation — Controlled group receives CIMT with baseline rehabilitation. Only receives CIMT without Robotic Gloves. Additional assessments may be conducted after 3 or 6 months to measure long-term effects.
  Arms: Group B

SUMMARY:
This study investigates the impact of CIMT, with and without robotic gloves, on hand dexterity and grip strength in children with hemiplegic CP, aiming to enhance motor skills and promote independence in daily activities. Conducted as a randomized controlled trial at DHQ Hospital, Mandi Bahauddin, the study involves two groups of children aged 6-12 with hemiplegic CP. One group of 17 children will receive CIMT alone with standard treatment, while the other 17 will receive CIMT combined with robotic glove assistance. The robotic glove device aids in flexion, extension, and individual finger movements, providing support for both isolated and coordinated finger actions. Each therapy session will last six hours and be held three to five days a week over four to eight weeks.

DETAILED DESCRIPTION:
Hemiplegic cerebral palsy (CP) often affects one side of the body, limiting functional abilities. Constraint-Induced Movement Therapy (CIMT) is a common intervention where the unaffected hand is restricted to encourage the use of the affected hand. Recently, the addition of robotic gloves has been proposed to improve outcomes, as they offer mechanical support and feedback to the affected hand. This study investigates the impact of CIMT, with and without robotic gloves, on hand dexterity and grip strength in children with hemiplegic CP, aiming to enhance motor skills and promote independence in daily activities. Conducted as a randomized controlled trial at DHQ Hospital, Mandi Bahauddin, the study involves two groups of children aged 6-12 with hemiplegic CP. One group of 17 children will receive CIMT alone with standard treatment, while the other 17 will receive CIMT combined with robotic glove assistance. The robotic glove device aids in flexion, extension, and individual finger movements, providing support for both isolated and coordinated finger actions. Each therapy session will last six hours and be held three to five days a week over four to eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years with Hemiplegic CP.
* Both Genders will be included.
* Fulfilling the CIMT criteria i.e. Up to 20 Degree Wrist Extension, up to 10 Degree
* Thumb Abduction and Up to 10 Degree Finger Extension.
* GMFCS level of 1 and 2.
* MAC Grade 2 and 3.
* Ability to understand and follow simple instructions.

Exclusion Criteria:

* Severe cognitive impairment or intellectual disability.
* Presence of other neurological disorders such as epilepsy.
* Children currently participating in other intensive physical therapy programs.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Grip Strength Test | 4-8 weeks
  The grip strength test and pinch strength is used to assess function of the hand using dynamometer. Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength
Box and Block Test | 4-8 weeks
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. The BBT is composed of a wooden box divided in two EFFECTS OF CIMT WITH AND WITHOUT ROBOTIC GLOVES IN CHILDREN WITH HEMIPLEGIC CP 11 compartments by a partition and 150 blocks. The BBT administration consists of asking the client to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Aftab Ansar Lodhi, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osuagwu BAC, Timms S, Peachment R, Dowie S, Thrussell H, Cross S, Shirley R, Segura-Fragoso A, Taylor J. Home-based rehabilitation using a soft robotic hand glove device leads to improvement in hand function in people with chronic spinal cord injury:a pilot study. J Neuroeng Rehabil. 2020 Mar 5;17(1):40. doi: 10.1186/s12984-020-00660-y. PMID 32138780